CLINICAL TRIAL: NCT03896633
Title: A BIOEQUIVALENCE STUDY OF THE GENERIC BRINZOLAMIDE 1% OPHTHALMIC SUSPENSION COMPARED TO REFERENCE LISTED DRUG AZOPT® (BRINZOLAMIDE) OPHTHALMIC SUSPENSION 1% IN SUBJECTS WITH PRIMARY OPEN ANGLE GLAUCOMA OR OCULAR HYPERTENSION
Brief Title: Therapeutic Equivalence Study of Generic Brinzolamide vs Azopt
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 883
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Results first posted 2021-06-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2021-05

CONDITIONS: Glaucoma; Open Angle or Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — brinzolamide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azopt 1% ophthalmic suspension (Active Comparator): Ophthalmic suspension
  Interventions: Drug: Azopt 1%
- Brinzolamide 1% ophthalmic suspension (Experimental): ophthalmic suspension
  Interventions: Drug: brinzolamide 1% ophthalmic suspension

INTERVENTIONS:
Drug: brinzolamide 1% ophthalmic suspension — brinzolamide 1% ophthalmic suspension
  Other Names: brinzolamide
  Arms: Brinzolamide 1% ophthalmic suspension
Drug: Azopt 1% — Azopt 1%, RLD
  Other Names: brinzolamide
  Arms: Azopt 1% ophthalmic suspension

SUMMARY:
The main purpose of this prospective study is to demonstrate the therapeutic equivalence of topical brinzolamide compared with AzoptTM

DETAILED DESCRIPTION:
The main purpose of this prospective study is to demonstrate the therapeutic equivalence of topical brinzolamide dosed three times daily compared with AzoptTM (brinzolamide ophthalmic suspension 1%) dosed three times daily in IOP reduction in patients with POAG or OH.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 18 years of age or older,
* diagnosed with primary open-angle glaucoma or ocular hypertension.

Exclusion Criteria:

* Patients with any form of glaucoma (such as secondary, congenital, juvenile or normal tension glaucoma, angle closure glaucoma) in either eye other than primary open-angle glaucoma,
* ocular hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 637 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2018-11-17 (Actual); Study Completion 2018-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Various, Bridgewater, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brinzolamide 1% Ophthalmic Suspension | Azopt 1% Ophthalmic Suspension
Started | 321 | 316
Completed | 312 | 306
Not Completed | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brinzolamide 1% Ophthalmic Suspension | Azopt 1% Ophthalmic Suspension | Total
Number analyzed (Participants) | 321 | 316 | 637
Age, Continuous [Mean (Full Range); unit: years] | 65.1 [20 to 91] | 63.8 [20 to 90] | 64.4 [20 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 190 | 389
  Male | 122 | 126 | 248
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 12 | 9 | 21
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 87 | 81 | 168
  White | 220 | 223 | 443
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP)
Time Frame: 6 weeks
Population: The Per Protocol Population was utilized for the primary outcome, included all randomized participants who met all inclusion/exclusion criteria, instilled 75% to 125% of the planned doses for the entire duration of the study, as verified by diaries, and who did not miss the scheduled applications for more than 3 consecutive days, and completed evaluations at Day 14 and Day 42 within the designated visit window (± 4 days) with no protocol deviations that would affect the treatment evaluation.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Brinzolamide 1% Ophthalmic Suspension | Azopt 1% Ophthalmic Suspension
Number analyzed (Participants) | 292 | 296
mmHg | 20.07 (3.269) | 19.89 (3.183)

2. Other Pre Specified Outcome: Change in Intraocular Pressure (IOP)
Description: Change in intraocular pressure (IOP) from baseline (Eligibility Visit 2) and after treatment.
Time Frame: 6 weeks
Population: The Per Protocol Population was utilized for this outcome; included all randomized participants who met all inclusion/exclusion criteria, instilled 75% to 125% of the planned doses for the entire duration of the study, as verified by diaries, and who did not miss the scheduled applications for more than 3 consecutive days, and completed evaluations at Day 14 and Day 42 within the designated visit window (± 4 days) with no protocol deviations that would affect the treatment evaluation.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Brinzolamide 1% Ophthalmic Suspension | Azopt 1% Ophthalmic Suspension
Number analyzed (Participants) | 292 | 296
mmHg | -4.85 (2.792) | -4.70 (2.861)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: One Brinzolamide participant did not receive treatment and is not included in the participant counts for safety. Two Brinzolamide participants received at least one dose of Azopt in error, and therefore the Azopt group has 2 additional participants for safety.
Arm/Group | Brinzolamide 1% Ophthalmic Suspension | Azopt 1% Ophthalmic Suspension
All-Cause Mortality (participants affected / at risk) | 0/320 | 0/318
Serious Adverse Events (participants affected / at risk) | 0/320 | 2/318
Other Adverse Events (participants affected / at risk) | 15/320 | 22/318
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brinzolamide 1% Ophthalmic Suspension (N=320) | Azopt 1% Ophthalmic Suspension (N=318)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brinzolamide 1% Ophthalmic Suspension (N=320) | Azopt 1% Ophthalmic Suspension (N=318)
Dysgeusia (Nervous system disorders) | 15 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/33/NCT03896633/Prot_SAP_000.pdf